CLINICAL TRIAL: NCT04385654
Title: Toripalimab Combined With Axitinib as Neoadjuvant Therapy for Advanced/Metastatic Non-clear Cell Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Hao Zeng, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TORAXI
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Neoadjuvant Therapy; Advanced Cancer; Metastatic Kidney Cancer
Keywords: Toripalimab; Axitinib; Neoadjuvant; Advanced/Metastatic; Non-clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis | interventions — toripalimab; spartalizumab; Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant toripalimab plus axitinib (Experimental): Toripalimab (240 mg,ivgtt,q3w) combined with Axitinib (5 mg,po,bid) was treated for 6 weeks and underwent surgery within 2-4 weeks
  Interventions: Drug: Toripalimab; Drug: Axitinib

INTERVENTIONS:
Drug: Toripalimab — Toripalimab (240 mg,ivgtt,q3w) was administered to patients for 6 weeks and underwent surgery within 2-4 weeks
  Other Names: anti-PD-1 antibody
Drug: Axitinib — Axitinib (5 mg,po,qd) was administered to patients for 6 weeks and underwent surgery within 2-4 weeks
  Other Names: TKIs

SUMMARY:
This is a single-arm phase II clinical trial to evaluate the initial efficacy and safety of toripalimab combined with axitinib as neoadjuvant therapy for advanced/metastatic non-clear cell renal cell carcinoma

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is a malignant tumor with a wide range of heterogeneity, including heterogeneous histological types. In addition to the most common clear cell carcinoma subtype (more than 80%), the remaining histological types are collectively referred to as non clear cell carcinoma (non-ccRCC), including papillary renal cell carcinoma (10-15%), chromophobe renal cell carcinoma (5%), and more rare Xp11.2 translocated RCC, unclassified as well as collecting duct carcinoma.

Recent advances in molecular immunology have promoted the discovery of immune checkpoint inhibitors (ICIs) and have been successfully applied in clinic. Blockade to programmed death receptor 1(PD-1) improves survival in patients with metastatic renal cell carcinoma (mRCC), but has not been validated in advanced RCC, especially immune combination TKIs drugs. Preoperative immunotherapy (IO) with immune plus TKIs, that is, neoadjuvant IO plus TKIs therapy, is of therapeutic value. Because primary tumors can serve as antigens for tumor-specific T cell activation, diffusion, and spread, and then activate immune system to monitor micrometastasis. Moreover, peripheral blood can be obtained during neoadjuvant therapy, which lays a foundation for the study of the in vivo effects of PD-1 inhibitors combined with TKIs on the microenvironment of primary tumors.

This study intends to validate the safety and feasibility of neoadjuvant immunotherapy combined to TKIs in patients with locally advanced/metastatic renal cell carcinoma. At the same time, this study intends to assess the relationship between somatic gene expression profiles and pathological responses, as well as the dynamic changes in the microenvironment, intratumoral, and immune biomarkers of primary renal cell carcinoma induced by immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1) age ≥18,<75; 2) histopathological evidence of renal cell carcinoma , histological type is non-clear cell renal cell carcinoma, and meet one of the following conditions :(1) clinical T stage ≥2, or lymph node positive, or nuclear grading ≥3; (2) confirmed by imaging or pathology that distant metastasis has occurred; 3) sections with formalin-fixed paraffin blocks or at least 10 um of tissue tumor biopsy samples for biomarker exploration studies; 4) ECOG score ≤1; 5) life expectancy above 6 months; 6) sign informed consent, and be able to follow the visit and related procedures stipulated in the program; 7) agree to collect tumor tissue, blood and other specimens required by this study and apply them to relevant studies; 8)important organs and bone marrow functions meet the following requirements: absolute neutrophil count (ANC) ≥1.5×109/L, platelet (PLT) ≥100×109/L, hemoglobin (HGB) ≥9g/dL;Liver function: serum total bilirubin (TBIL) ≤1.5 times normal upper limit (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5 times ULN, serum albumin (ALB) ≥ 2.8g /dL. Renal function: serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥40 mL/min; 9) cardiac function met the following conditions: baseline electrocardiogram (ECG) had no evidence of PR prolongation or AV block;

Exclusion Criteria:

* 1) patients with other malignant tumors with different primary sites or histology from the tumor evaluated in this study within 2 years of personal history, except those with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or cervical carcinoma in situ under good control; 2) major surgery or severe trauma within 4 weeks before enrollment; 3) immunosuppressive drugs were used within 4 weeks prior to the first dose of study therapy, excluding local glucocorticoids, inhaled or otherwise, or systemic glucocorticoids at physiological doses (i.e., no more than 10mg/ d prednisone or equivalent doses of other glucocorticoids); 4) known or suspected active autoimmune diseases (congenital or acquired), such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroiditis, etc. Patients with type 1 diabetes with good insulin control can also be enrolled.

  5) known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation; 6) allergic to any component of monoclonal antibody; 7) suffering from other uncontrolled serious diseases, including but not limited to: A) severe infection in the active phase or clinically poorly controlled; B) HIV infection (HIV antibody positive); C) acute or chronic active hepatitis b (HBsAg positive and HBV DNA>1*103/ml) or acute or chronic active hepatitis c (HCV antibody positive and HCV RNA>15IU/ml); D) active tuberculosis, etc.; 8) class iii-iv congestive heart failure (New York heart association classification), poorly controlled and clinically significant arrhythmia; 9) uncontrolled arterial hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg); 10) had any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, etc. within 6 months before the selected treatment; 11) diseases requiring the use of warfarin (coumarin) for anticoagulant treatment; 12) uncontrolled hypercalcemia (more than 1.5 mmol/L of calcium or calcium greater than 12 mg/dL or adjusted serum calcium greater than ULN), or symptomatic hypercalcemia requiring continued bisphosphate treatment; 13) accompanied by other malignant tumors (except those that have been cured, such as cervical carcinoma in situ, non-melanoma skin cancer, etc.); 14) other acute or chronic diseases, psychiatric disorders, or laboratory abnormalities that may result in increased risk associated with study participation or study drug administration, or interference with the interpretation of study results, and ineligibility to participate in the study as determined by the investigator; 15) pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response (MPR) | 6 week
  The residual tumor cells (% RVT) were calculated according to immune related pathologic response criteria (irPRC), MPR is defined as %RVT<10%
Pathologic Complete Response (pCR) | 6 week
  The residual tumor cells (% RVT) were calculated according to immune related pathologic response criteria (irPRC), pCR is defined as %RVT<0%
Pathologic No Response (pNR) | 6 week
  The residual tumor cells (% RVT) were calculated according to immune related pathologic response criteria (irPRC), pCR is defined as %RVT>90%

SECONDARY OUTCOMES:
Objective response rate (ORR) | 6 week
  Rate of patients achieving a complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) and immune-related response criteria (IRC)
Disease-free survival(DFS) | Up to 24 months
  DFS is defined as the time from treatment to recurrence of tumor or death
Progression-free survival(PFS) | Up to 24 months
  PFS is defined as the time from treatment to progression disease or death. Progression disease is assessed by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) and immune-related response criteria (IRC)
Overall survival(OS) | Up to 24 months
  OS is defined as the time from treatment to death.
Functional Assessment of Cancer Therapy (FACT)-Kidney Symptom Index 19 (FKSI-19) | Up to 24 months
  FKSI-19 score change over time from baseline to disease progression. The scale of FKSI-19 is from 0 to 48, and higher scores indicate worse quality of life.
Functional Assessment of Cancer Therapy- Kidney Symptom Index- Disease related Symptoms (FKSI-DRS) | Up to 24 months
  FKSI-DRS score change over time from baseline to disease progression. The scale of FKSI-DRS is from 0-36, and higher scores indicate worse quality of life.
EuroQol five-dimension scale (EQ-5D) | Up to 24 months
  EQ-5D-5L score change over time from baseline to disease progression. The EQ-5D-5L is consisted of five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Higher scores indicate poorer health.
Visual analogue scale (VAS) | Up to 24 months
  VAS pain score change over time from baseline to disease progression. The scale of VAS is from 0-10, and higher scores indicate worse symptom of pain.
Frequency of treatment-related adverse events (AEs) | Up to 24 months
  Treatment related adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Perioperative complication rate | From surgery to postoperative 3 months
  Perioperative complications assessed by The Clavien-Dindo Classification

IPD SHARING:
Plan to Share IPD: No